CLINICAL TRIAL: NCT03483610
Title: Piloting Interventions to Improve Adherence to Cervical Cancer Screening Recommendations Among Emergency Department Patients
Brief Title: Promoting Cervical Cancer Screening for Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Adler, Associate Professor of Emergency Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSRB00070962
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- screening and referral (Active Comparator)
  Interventions: Behavioral: Provider Referral
- behavioral intervention (Active Comparator)
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Provider Referral — Participants will be asked if they are up-to-date on their cervical cancer screening. If not they will be referred to a provider. At the end of the study they will receive a 10 minute follow up telephone survey to collect data screening status and views on cervical cancer screening.
  Arms: screening and referral
Behavioral: Text Messaging — Participants will be asked if they are up-to-date on their cervical cancer screening. If not they will be referred to a provider. They will also receive a total of 3 text messages at 30-day intervals encouraging follow-up for cervical cancer screening. They will receive a 10 minute follow up telephone survey to collect data screening status and views on cervical cancer screening.
  Arms: behavioral intervention

SUMMARY:
The purpose of this study is to learn methods to encourage women to get recommended cervical cancer screening. Cervical cancer screening is an important part of cervical cancer prevention. The study team will determine if the patient is currently up-to-date with cervical cancer screening recommendations. If the patient is not up-to-date, then they will be randomly assigned to one of two interventions. One intervention consists only of referral to a women's health care provider to obtain cervical cancer screening. The other intervention consists of receiving a total of 3 text messages at 30-day intervals encouraging follow-up for cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient in the Emergency Department of the University of Rochester Medical Center
* Women
* Age 21 - 65

Exclusion Criteria:

* Past hysterectomy with cervical removal
* Known infection with HIV (screening recommendations for women with HIV differ from the general population)
* Non-English speaking
* Inability to consent
* Lack of text-capable mobile phone and/or inability to use text function

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women get cervical cancer screening
Enrollment: 95 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Department of Emergency Medicine, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Withing one year of publication

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All enrollment occurred over an 8 week period (June-August 2018) at a large (approximately 118,000 annual patient visits), urban, academic ED. Eligible patients were female, ages 21-65 years, and demonstrating decisional capacity to consent to participate.
Pre-assignment Details: Women with past hysterectomy with cervical removal, known HIV infection, inability to consent, non-English speaking, or not having a text-capable phone were excluded. 502 eligible approached to achieve the target of 450. The primary reason for declining was lack of interest. Among consented potential-participants, 355 (79%) were adherent with screening recommendations and their participation ended. The remaining 95 participants that were determined to be eligible to be randomized.
Period: Overall Study
Arm/Group | Screening and Referral | Behavioral Intervention
Started | 47 | 48
Completed | 28 | 21
Not Completed | 19 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening and Referral | Behavioral Intervention | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 48 | 95
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 39 | 39 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 27 | 24 | 51
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Scheduled or Completed Cervical Cancer Screening
Time Frame: 150 days
Measure: Count of Participants; unit: Participants
Arm/Group | Screening and Referral | Behavioral Intervention
Number analyzed (Participants) | 28 | 21
Participants | 28 | 21

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected for participants during their 150 days of participation
Description: The study was strictly focused on survey methods & text to receive cervical cancer screening. The primary risk of this study was breach of confidentiality. No SAE's were reasonably expected to occur from a study of this nature. Additionally, the follow-up period was also 150 days.
Arm/Group | Screening and Referral | Behavioral Intervention
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 0/47 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT03483610/Prot_SAP_000.pdf